CLINICAL TRIAL: NCT06513663
Title: Exercise as Maintenance Therapy in Advanced Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tarah J Ballinger, MD, Assistant Professor of Clinical Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CTO-IUSCCC-0865
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer; Non Small Cell Lung Cancer; Metastatic Lung Cancer
Keywords: lung cancer; exercise; non small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Intervention (Experimental): Eligible and consented participants randomized to the exercise arm will work with an exercise trainer three times weekly for 12 weeks. Training sessions will be delivered virtually using HIPPA Complaint IU Health Zoom. These sessions will last 60 minutes and include cardiovascular exercise, resistance training, and balance or stretching exercise. The participants will be able to use any equipment they already have at home but will be provided a heart monitor and a set of resistance bands.
  All sessions will have a moderate-intensity training goal, defined as 40-80% of heart rate reserve (HRR). Cardiovascular exercise will include any at-home equipment available to the participants or follow a Tabata-style program. Resistance training will include a full body workout, emphasizing all major muscle groups. Trainers will progress or regress intensity levels based on the participant's rate of perceived exertion (RPE), heart rate, and individual response during each session.
  Interventions: Behavioral: Exercise Intervention
- Usual Care (No Intervention): Participants randomized to usual care arm will receive care per their treatment team. Usual care participants are encouraged to exercise but will not be provided components of the intervention. Participants in the usual care arm will be given usual care handouts at baseline.

INTERVENTIONS:
Behavioral: Exercise Intervention — Eligible and consented participants randomized to the exercise arm will work with an exercise trainer three times weekly for 12 weeks. Training sessions will be delivered virtually using HIPPA Complaint IU Health Zoom. These sessions will last 60 minutes and include cardiovascular exercise, resistance training, and balance or stretching exercise. The participants will be able to use any equipment they already have at home but will be provided a heart monitor and a set of resistance bands.
  All sessions will have a moderate-intensity training goal, defined as 40-80% of heart rate reserve (HRR). Cardiovascular exercise will include any at-home equipment available to the participants or follow a Tabata-style program. Resistance training will include a full body workout, emphasizing all major muscle groups. Trainers will progress or regress intensity levels based on the participant's rate of perceived exertion (RPE), heart rate, and individual response during each session.
  Arms: Exercise Intervention

SUMMARY:
The purpose of this study is to examine how a multimodality (having or using a variety of methods to do something) exercise intervention may improve survival, function, and quality of life in participants with advanced lung cancer.

DETAILED DESCRIPTION:
This study is a randomized control trial at a single institution comparing advanced lung cancer patients undergoing supervised home-based exercise program versus usual care. The intervention is a supervised home-based exercise program that will be coordinated by the MOVE program. The regimen will be 12 weeks in duration, three times a week, and administered by a trained professional virtually.

Participants will be randomized 1:1 to the exercise or usual care arm. Participants will be stratified on baseline frailty by the SPPB.

Primary Objective To compare changes patient-reported fatigue (by FACT-F survey) from baseline to post-intervention in patients with locally advanced and advanced lung cancer receiving maintenance immunotherapy undergoing a supervised home-based exercise program versus usual care.

Secondary Objectives

1. To compare changes in cardiorespiratory fitness measured by VO2peak, estimated as time on the treadmill during ramp treadmill test, from baseline to post-intervention in patients with locally advanced/advanced lung cancer receiving maintenance immunotherapy undergoing a supervised home-based exercise program versus usual care.
2. To compare changes in physical function measured by the short physical performance battery from baseline to post-intervention in patients with locally advanced/advanced lung cancer receiving maintenance immunotherapy undergoing a supervised home-based exercise program versus usual care.
3. To compare changes in muscle mass and muscle density measured on CT scans for disease monitoring and bioimpedance analysis from baseline to post-intervention in patients with locally advanced/advanced lung cancer receiving maintenance immunotherapy undergoing a supervised home-based exercise program versus usual care.
4. To compare changes in depression scores by HADS survey from baseline to post-intervention in patients with locally advanced and/or advanced lung cancer receiving maintenance immunotherapy undergoing a supervised home-based exercise program versus usual care.
5. To compare the proportion of patients who are "fatigued," defined as a FACT-F score of <43 at post-intervention between the exercise and usual care arms.
6. To evaluate uptake and adherence of supervised home-based exercise program in patients with locally advanced and/or advanced lung cancer receiving maintenance immunotherapy or targeted therapy, measured by the percentage of patients who consented to the study and percentage of training sessions attended by patients in the exercise arm.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Known diagnosis of locally advanced (stage III) or metastatic NSCLC
3. Patient is currently receiving maintenance immunotherapy for at least 1 month and planned for at least 3 additional months of therapy

   1. Patients receiving maintenance therapy refers to patients with stable disease or partial response to therapy, including patients who have had a history of disease progression but are currently stable or responding to a different therapy
   2. Patients previously receiving chemotherapy are eligible as long as at least one month has elapsed since completing chemotherapy. Those currently receiving chemotherapy are not eligible.
4. Patient is willing and able to participate in a supervised home-based exercise program as determined by the MOVE program

   a.Participants must have internet access and equipment to participate in virtual exercise
5. ECOG performance status of 0-2

Exclusion Criteria:

1. Already meeting exercise guidelines and participating in at least 150 minutes of moderate or vigorous exercise per IPAQ
2. Unable to participate in the supervised home-based exercise program as determined by the MOVE program
3. Medical co-morbidities that preclude patient from participating in supervised exercise, including but not limited to:

   * Advanced heart failure
   * Advanced respiratory disease requiring home oxygen use
   * Uncontrolled psychiatric disorders
   * History of fragility fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in patient-reported fatigue | baseline, week 12, and week 24
  Measured by Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) survey

SECONDARY OUTCOMES:
Change in cardiorespiratory fitness | baseline, week 12, and week 24
  Measured by VO2peak, estimated as time on the treadmill
Change in physical performance battery | baseline, week 12, and week 24
  total score on short physical performance battery
Change in muscle mass | baseline, and week 12
  measured by mg/kg2 on HU on CT scans
Change in muscle density | baseline, and week 12
  measured by mg/kg2 on HU on CT scans
Change in depression | baseline, week 12, and week 24
  measured by total score of HADS survey
Proportion of patients who are "fatigued" | baseline, week 12, and week 24
  measured by FACT-F score of <43
Uptake of the study | date open to accrual until closed to accrual, up to 5 years
  the proportion of total patients approached, screened, and ultimately completing the baseline assessments
Adherence with the intervention defined | baseline to post 12-week intervention
  the proportion of scheduled sessions attended by participants randomized to the exercise intervention arm

CONTACTS AND LOCATIONS:
Overall Officials: Tarah J Ballinger, MD, Principal Investigator — Indiana University
Locations (3):
- United States (3):
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Indiana University Melvin & Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana